CLINICAL TRIAL: NCT01103050
Title: A Randomized, Double-blind, Double-dummy, Placebo Controlled Three-period Incomplete Cross Over Study to Compare the Effect of Combined Treatment With QAV680 and Cetirizine on Total Nasal Symptom Score in Allergic Rhinitis Patients in an Environmental Exposure Chamber
Brief Title: A Cross Over Study to Compare the Effect of Combined Treatment With QAV680 and Cetirizine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAV680A2204
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic inflammation; Seasonal rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- QAV680 + Cetirizine Placebo (Active Comparator)
  Interventions: Drug: QAV680 + Cetirizine Placebo
- QAV680 + Cetirizine (Experimental)
  Interventions: Drug: QAV680 + Cetirizine
- Cetirizine + QAV680 Placebo (Active Comparator)
  Interventions: Drug: Cetirizine + QAV680 Placebo
- QAV680 Placebo + Cetirizine Placebo (Placebo Comparator)
  Interventions: Drug: QAV680 Placebo + Cetirizine Placebo

INTERVENTIONS:
Drug: QAV680 + Cetirizine Placebo
  Arms: QAV680 + Cetirizine Placebo
Drug: QAV680 + Cetirizine
  Arms: QAV680 + Cetirizine
Drug: Cetirizine + QAV680 Placebo
  Arms: Cetirizine + QAV680 Placebo
Drug: QAV680 Placebo + Cetirizine Placebo
  Arms: QAV680 Placebo + Cetirizine Placebo

SUMMARY:
This study will determine the capacity of more frequent dosing of QAV680 to suppress allergic inflammation. The study will investigate the paradigm of multiple receptor antagonism in allergic disease by combining QAV680 with a second generation H1 histamine receptor antagonist to assess possible additive or synergistic anti-allergic effects of the two compound classes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical history of intermittent allergic rhinitis with seasonal onset and offset of nasal allergy symptoms during each of the last two ragweed allergy seasons
* positive skin prick test to ragweed allergen within twelve months of screening

Exclusion criteria:

* Use of any medication used to treat allergy (administered via any route), such as: pseudoephedrine, antihistamines, ipratropium bromide, cromoglycates, corticosteroids, immunotherapy or other antiinflammatory or immunosuppressive agents, or any other medication administered via the nasal or ocular routes)
* Within the last three years a recurrent history of acute or chronic bronchospastic disease including moderate-severe asthma or chronic obstructive pulmonary disease
* Nasal conditions such as nasal septal perforations,nasal polyps, sinus disease, chronic nasal obstruction

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2010-07-28 (Actual); Study Completion 2010-07-28 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score measured during allergen exposure | 14 Days

SECONDARY OUTCOMES:
Nasal airway patency assessed by acoustic rhinometry during allergen exposure | 14 days
Nasal secretion weight during allergen exposure | 14 days
Total Nasal Symptom Score & Total Ocular Symptom Score measured during allergen exposure | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Ontario, Canada

REFERENCES:
- See also: Publication Link QAV680, cetirizine and their combination reduce nasal symptoms in patients with intermittent allergic rhinitis in an environmental exposure chamber — http://www.ers-education.org/home/browse-all-content.aspx?idParent=136559